CLINICAL TRIAL: NCT03486639
Title: Urodynamics and Clinical Factors That Are Associated With Bladder Over-sensitivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Kobi Stav, Head of the Neuro-Urologic Unit, Assaf-Harofeh Medical Center
Other Study IDs: 0101-17-ASF
Record Dates: First submitted 2018-03-24; First posted 2018-04-03 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Overactive Bladder Syndrome; Bladder Outlet Obstruction; Benign Prostate Enlargement; Stress Incontinence (Female) (Male); Bladder Disease
Keywords: Urodynamics; Bladder sensation; confounding factors
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Prostatic Hyperplasia; Urinary Incontinence, Stress; Urinary Bladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing urodynamic: All patients older than 18 who are refered for Urodynamics examination
  Interventions: Other: IPSS questionnaire

INTERVENTIONS:
Other: IPSS questionnaire — IPSS is an 8 question (7 symptom questions + 1 quality of life question) written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of patients with lower urinary tract symptoms. It was validated for both genders.
  Other Names: International Prostate Symptoms Score

SUMMARY:
Urodynamic examination evaluates storage and empting phases of the urinary bladder. It enables the clinician to correlate physiologic findings to patients' complains. The data gathered during the examination divided to storage and empting.

During the storage phase, bladder sensation is measured while the bladder is filled with sterile water. During years of practice, we noticed that early sensation (bladder over-sensitivity) is occasionally associated with bladder outlet obstruction (as demonstrated in the emptying phase of the examination.

DETAILED DESCRIPTION:
The study includes patients who were referred to Urodynamics examination due to lower urinary tract symptoms. There is no actual intervention during the examination. Though, patients are asked to fill an International prostate symptom score (IPSS-questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* All patients refered to Asaf HaRofeh Medical Center for Urodynamic examination

Exclusion Criteria:

* Inability to sign an informed concent
* Administration of analgesics 8 hours prior to the examination
* Known urethral stricture
* Chronic bladder or urethral pain
* Active cystitis
* Permanent urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients reffered to Asaf HaRofeh Medical Center for Urodynamic examination
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-19 (Estimated)

PRIMARY OUTCOMES:
Early sensation during the filling phase | During the urodynamic examination
  Bladder oversensitivity (early sensation), a diagnosis made by symptoms and urodynamic investigations. Defined as an increased perceived bladder sensation during bladder filling with specific cystometric findings of: (i) an early first desire to void; (ii) an early strong desire to void, which occurs at low bladder volume; (iii) a low maximum cystometric bladder capacity; no abnormal increases in detrusor pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofe Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No
No plans of sharing participants data

REFERENCES:
- [Background] Campbell Walsh Urology chapter 73
- [Background] Lee WC, Wu HP, Tai TY, Yu HJ, Chiang PH. Investigation of urodynamic characteristics and bladder sensory function in the early stages of diabetic bladder dysfunction in women with type 2 diabetes. J Urol. 2009 Jan;181(1):198-203. doi: 10.1016/j.juro.2008.09.021. Epub 2008 Nov 14. PMID 19013605
- [Background] Schurch B, Schmid DM, Kaegi K. Value of sensory examination in predicting bladder function in patients with T12-L1 fractures and spinal cord injury. Arch Phys Med Rehabil. 2003 Jan;84(1):83-9. doi: 10.1053/apmr.2003.50007. PMID 12589626
- [Background] El-Zawahry A, Alanee S, Malan-Elzawahry A. The Use of Urodynamics Assessment Before the Surgical Treatment of BPH. Curr Urol Rep. 2016 Oct;17(10):73. doi: 10.1007/s11934-016-0626-y. PMID 27535043